CLINICAL TRIAL: NCT01137669
Title: Phase I Trial of ZOSTAVAX® Prior to Renal Transplantation
Brief Title: ZOSTAVAX® in Renal Transplant Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 09-0016
Record Dates: First submitted 2010-06-03; First posted 2010-06-04 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2015-10

CONDITIONS: Herpes Zoster
Keywords: immunocompromised,parent protocol,shingles,varicella-zoster virus,ZOSTAVAX®
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator): 10 subjects to receive placebo subcutaneously.
  Interventions: Other: Placebo
- ZOSTAVAX® (Experimental): 30 subjects to receive 0.65 mL ZOSTAVAX® subcutaneously.
  Interventions: Biological: Live attenuated herpes zoster vaccine

INTERVENTIONS:
Biological: Live attenuated herpes zoster vaccine — ZOSTAVAX® (Zoster Vaccine Live) is a live attenuated vaccine provided as a single-dose, sterile, lyophilized, preservative-free frozen formulation. The vaccine will be supplied in 3-mL glass vials. Sterile diluent will be used to reconstitute study vaccine. The reconstituted vial will be gently agitated to mix thoroughly. The entire contents of the reconstituted vaccine vial (approximately 0.65 mL) will be withdrawn into a syringe. The vaccine will be administered immediately subcutaneously in the deltoid region.
  Arms: ZOSTAVAX®
Other: Placebo — Placebo for Zoster Vaccine Live (ZOSTAVAX®) is sterile normal saline which will be obtained from the Fisher Repository in single-dose containers. 0.9% Sodium Chloride Injection, USP is a sterile, nonpyrogenic, isotonic solution of sodium chloride and water for injection. The placebo will be administered subcutaneously in the deltoid region.
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the safety of a licensed zoster vaccine, ZOSTAVAX® (Zoster Vaccine Live) in 40 subjects, age 18 years or older, with chronic kidney disease (CKD) who are scheduled to receive a living donor kidney transplant. ZOSTAVAX® is not licensed for use in immunosuppressed persons and in the United States for individuals less than 50 years of age. Subjects will receive either ZOSTAVAX® vaccine or placebo (inactive substance) no less than 4 weeks prior to their kidney transplant. Study procedures include: physical exam, blood samples and documentation of daily temperatures and/or side effects in a diary following vaccination. Participants may be involved in study related procedures for up to 18 months.

DETAILED DESCRIPTION:
Infection with varicella-zoster virus (VZV) produces a life-long latent infection in sensory ganglia. Reactivation of viral replication from latency results in a number of clinical syndromes, most commonly herpes zoster, or shingles. Herpes zoster is typically a unilateral vesicular rash in a dermatomal distribution accompanied by radicular pain that may be severe. Immunocompromised persons are at higher risk for herpes zoster than immunocompetent adults. The markedly increased risk of herpes zoster in organ transplant recipients suggests that this population would benefit substantially if a similar strategy could be adopted. The currently licensed zoster vaccine, ZOSTAVAX® (Zoster Vaccine Live), is not licensed for use in immunosuppressed persons and in the United States for those less than 50 years of age. A small Phase I study is important to address immunogenicity in patients with Chronic Kidney Disease (CKD) prior to transplantation as well as safety and persistence of immune responses following transplantation. This study is a multi-center, double blind, randomized, placebo-controlled trial of ZOSTAVAX® immunization in subjects who will undergo renal transplantation from a living donor or are wait-listed for a deceased donor no less than 4 weeks prior to transplantation. The primary objective of this study is to assess the safety of ZOSTAVAX® when administered to subjects with CKD a minimum of 4 weeks prior to live donor renal transplantation. This will be accomplished by comparing the rates of specific local and systemic reactogenicity events and adverse events (AEs) between the vaccine and placebo groups. Subjects likely to be suitable for renal transplant and who have an identified living donor will be consented for screening serology for antibodies to VZV if such serology is not standard of care or serostatus is not known. Subjects with positive VZV serology, an identified living donor, and meeting inclusion and exclusion criteria will provide signed informed consent for study enrollment. Subjects will be randomized to receive either active vaccine (ZOSTAVAX®) [30 subjects] or placebo vaccine [10 subjects]. Blood will be drawn on day 0 (day of vaccine) prior to vaccine administration for assessment of baseline humoral and cellular immunity to VZV. Subjects will receive ZOSTAVAX® or placebo vaccination. At approximately 5 weeks post-vaccination, subjects will have blood drawn for measurement of humoral and cellular immune response. Subjects will undergo living donor renal transplant with immunosuppression according to standard of care at each institution. All transplanted subjects will receive anti-viral prophylaxis for 3 months post-transplant, consisting of either valganciclovir (or ganciclovir) or acyclovir (or valacyclovir or famciclovir) depending on risk of cytomegalovirus (CMV) disease. Subjects will be followed and treated by the renal transplant team at each center according to local standard of care with concomitant monitoring by the vaccine study teams. Subjects will have blood drawn for humoral and cell-mediated immune assays at day 0, and week 5 post vaccination, and 6 months and 12 months post-transplantation if they undergo transplantation. Parent protocol to sub-study 09-0025.

ELIGIBILITY:
Inclusion Criteria:

-Subjects must be willing and able to provide informed consent prior to study procedures. -Age 18 years or older at the time of vaccination. -Chronic kidney disease (CKD) activated on the United Network for Organ Sharing (UNOS) deceased donor waitlist or anticipating living donor renal transplant no sooner than 4 weeks following vaccination. -Varicella Zoster Virus (VZV) seropositive by local laboratory or Center for Disease Control (CDC) serologic testing -Negative pregnancy test (women of childbearing age potential) performed at enrollment- or within 48 hours prior. The use of contraception for women of childbearing potential will be per renal transplant team's standard of care

Exclusion Criteria:

-Any pharmacologic immunosuppression at the time of enrollment, within one year prior to enrollment, or between enrollment and transplant (e.g., for underlying autoimmune disease or previous failed allograft). This includes prednisone at >/= 0.3 mg/kg/day or steroid equivalent for > 10 days, any use of anti-metabolites (azathioprine, mycophenolic acid, cytoxan), leflunomide, TNF-alpha inhibitors, calcineurin inhibitors, mTOR inhibitors, IL-6 or IL-6 receptor inhibitors. -Any transplant other than solitary kidney (e.g., no kidney/pancreas, kidney/liver transplants). Second kidney transplants are permitted. -Anticipated use of any post-transplant experimental immunosuppressive agent -Prior ZOSTAVAX® or Varivax® vaccination -Shingles or any other herpes zoster within 12 months of planned vaccination -Receipt of any killed vaccines within 2 weeks prior and 4 weeks following study vaccination or receipt of any live vaccines within 4 weeks prior and 6 weeks following study vaccination -Intercurrent illness at time of planned vaccination -Inability to vaccinate in either arm (e.g. due to A-V fistula or graft) -Known Human immunodeficiency virus (HIV) infection, Hepatitis C virus (HCV) infection, or chronic hepatitis B determined from review of laboratory data obtained from pre-transplant evaluation by renal transplant team. Note positive IgG hepatitis B surface antibody alone (negative HBcAb and negative IgM) is indicative of vaccine induced immunity and is not grounds for exclusion -History of anaphylactic/anaphylactoid reaction to gelatin, neomycin, or any other components of the vaccine -Asthma requiring systemic or inhaled steroid treatment within 12 months prior to enrollment -Allergy to ganciclovir, valgancyclovir, acyclovir, or famciclovir -Panel Reactive Antibody (PRA) >/= 20 percent or donor-specific sensitization (by solid phase assay or flow cytometry) or treatment with intravenous immunoglobulin (IVIG) for desensitization prior to transplant -History of primary or acquired immunodeficiency states. -Routine use of anti-viral prophylaxis for Herpes Simplex Virus (HSV) at the time of vaccination or within 3 months prior -Any other condition that in the opinion of the investigator might interfere with the subject's safety or ability to participate in the study -Abnormal screening laboratory data resulting in a disqualification of transplant candidacy. Abnormalities due to underlying disease (e.g., renal failure, anemia, hyperlipidemia, cardiovascular disease, diabetes) are not exclusionary except as denoted above for HIV, hepatitis B, hepatitis C, autoimmune disease. -The subject is currently participating in a study that involves an experimental agent (vaccine, drug, biologic, device, blood product, or medication) or has received an experimental agent within 1 month prior to enrollment in this study, or expects to receive another experimental agent during participation in this study. -The subject has a diagnosis of schizophrenia, bi-polar disease, or other severe (disabling) psychiatric diagnosis identified at the pre-transplant evaluation. -The subject has been hospitalized within the past 5 years prior to enrollment for psychiatric illness, history of suicide attempt or confinement for danger to self or others identified at the pre-transplant evaluation. -Dual listing at more than one transplant center. -Unwilling to be temporarily inactivated on UNOS wait list for 4 weeks post vaccination.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Biopsy proven graft rejection | During 12 months post- vaccination or post- transplantation
Safety: any occurrence of proven [polymerase chain reaction (PCR) confirmed] vaccine strain varicella zoster virus (VZV) infection at any site not contiguous with the injection site. | Entire post-immunization period up to 12 months following transplantation.
Safety: incidence of grade 3 or higher vaccine related adverse events (AEs) and vaccine related serious adverse events (SAEs). | During the 4 weeks post-immunization.
Safety: incidence of vaccine related serious adverse events (SAEs). | During 12 months post- vaccination or post-transplantation
Safety: increase of panel reactive antibody (PRA) by greater than or equal to 10% (e.g., from 10% to 20%) or newly positive donor specific cross match (DXM) after immunization in the absence of any other attributable cause. | Prior to vaccination, to following vaccination while on the wait list (for up to 12 months)
Safety: increase of panel reactive antibody (PRA) by greater than or equal to 10% (e.g., from 10% to 20%) or newly positive donor specific cross match (DXM) prior to transplantation in the absence of any other attributable cause. | Study Day 0, through Study Day 35 post vaccination, or to the time of transplantation in those subjects who are transplanted. The ideal time for transplantation is 6 weeks post vaccination.

SECONDARY OUTCOMES:
Immune response: changes from baseline glycoprotein-based enzyme-linked immunosorbent assay (gpELISA) varicella zoster virus (VZV) antibody titer. | Approximately 5 weeks post immunization, 6 months and 12 months post-vaccination or 6 months and 12 months post-transplantation.If transplantation occurs >12 weeks post-vaccination, a repeat pre-transplant baseline is optional.
Immune response: changes from baseline number of VZV specific T cells by flow cytometry measuring intracellular interleukin-2 (IL-2), interferon (IFN)-gamma, and tumor necrosis factor (TNF)-alpha after stimulation with VZV antigens. | Approximately 5 weeks post-immunization, 6 months and 12 months post-immunization or post-transplantation. If transplantation occurs >12 weeks post-vaccination, a repeat pre-transplant baseline is optional.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Iowa - Vaccine Research and Education Unit, Iowa City, Iowa
  - University of Maryland Baltimore - School of Medicine - Medicine, Baltimore, Maryland
  - Vanderbilt University - Medicine - Infectious Diseases, Nashville, Tennessee